CLINICAL TRIAL: NCT02925507
Title: Computerized Acoustic Swallowing Evaluation in Patients With Stroke
Brief Title: Computerized Acoustic Swallowing Evaluation
Acronym: CASE
Status: Withdrawn | Type: Observational
Why Stopped: Problems with biosensor not working properly and not functional for study
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Pamela Roberts, Director, Cedars-Sinai Medical Center
Other Study IDs: Pro00044374
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Deglutition Disorders; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Healthy patients with no neurologic impairments or disease
  Interventions: Other: Swallowing Screen
- Stroke Subjects: Patients with new onset stroke for ischemic, hemorrhagic or TIA
  Interventions: Other: Swallowing Screen

INTERVENTIONS:
Other: Swallowing Screen — Patient will be ask to undergo a swallowing screen by study staff

SUMMARY:
It is the purpose of this study to determine if a commercially available electronic stethoscope synchronized with an smart phone or iPad application can be used as an accurate and objective screening tool for measuring dysphagia. The investigators plan to do so in two phases; in Phase I the investigators will recruit normal subjects to establish normal swallowing patterns, as well as optimal sensor placement; and in Phase II the investigators will compare the recordings obtained by the electronic stethoscope with those obtained using videofluoroscopy.

DETAILED DESCRIPTION:
In this study, the investigators will use commercially available electronic stethoscope to assess dysphagia in patients who have recently experienced a stroke. The Eko Core electronic stethoscope is approved by the Food and Drug Agency (FDA) is currently available for use in the health care context.

Phase I

In the first phase of this study the investigators will try to establish the electronic stethoscope's measurements for normal swallowing patterns. The investigators will recruit healthy controls and auscultate for swallowing sounds at three locations: in the anterolateral section of the neck, in the posterior section of the neck, and in the superior sternum as illustrated in Figure 1. After the sensors are placed, participants will be asked to perform the following tests:

* Dry Swallow - ask participant to swallow their saliva
* Ask participant to swallow 1 teaspoon of water
* Ask participant to swallow 3 ounces of water (continuous)
* Ask participant to swallow one teaspoon of applesauce
* Ask participant to chew one cracker Healthy subjects will be recruited by advertisement using a flyer. Interested individuals will be able contact the study coordinator by email or phone. Subsequently, the participants will present for consenting and testing at the CSMC rehabilitation gym (North Tower 7215) or Pacific Theaters Building (116 N. Robertson) at a mutually agreed time.

The results of these tests will be used to determine the electronic stethoscope's measurements for a normal swallowing pattern.

Additionally, the investigators will determine optimal sensor location by measuring the quality of the recordings obtained in each location, and getting participant input with regarding their preferred sensor location. Signal quality will be determined by observing the loudness of the swallowing signal relative to the loudness of background noises (heartbeat, pulse, etc.) in each of the three locations.

Phase II As part of their standard of care, all stroke patients at CSMC undergo a swallowing screen by the nursing staff at bedside. If a patient fails the bedside screen, a referral is made to the physician for a clinical swallowing evaluation by a swallowing therapist. If the patient fails the clinical swallowing evaluation, the referral is made to the physician for an instrumental swallowing evaluation which is often the videofluoroscopy swallowing study. At bedside, the electronic stethoscope will be used to monitor the patients' pharyngeal acoustic signals while they undergo swallowing evaluations monitored by members of the research team.

During Phase II all subjects will undergo evaluation by the electronic stethoscope. Regarding VSS, it is entirely dependent upon the managing medical team and the physician.

The investigators anticipate that a number of patients will undergo VSS. If VSS is required, the order and timing will be determined by the medical team. Given the dynamic nature of the acute inpatient setting, details such as timing of VSS cannot be anticipated.

Potential participants will be identified through the daily stroke list on CS-Link, which is reviewed by the investigators who have access to this list as part of routine daily operations. The investigator has access to the patient list as part of quality oversight. Per request for waiver of consent/authorization, patients will be selected from this list based on inclusion/exclusion criteria. Subsequently, the treating physician will be contacted for approval to recruit the patient. Once approval is given, the investigator will then visit the patient and ask if he or she is willing to participate. The investigator will only consent patients that are able to communicate clear understanding of the study, by demonstrating that they understand purpose, procedure, risks and benefits of the study. If the patient cannot understand the purpose of the study, risks, and benefits they will not be consented.

Eligible patients will be approached by a member of the research team who will discuss the study in detail with them and obtain consent.

Once consent is obtained, the electronic stethoscope will be placed on the location found in Phase I to be optimal, and the patient will be asked to perform the following tests at bedside and during the videofluoroscopy swallowing study:

* Dry Swallow-Ask patient to swallow their saliva
* Ask patient to swallow 1 teaspoon of water
* Ask patient to swallow 3 ounces of water (continuous)
* Ask patient to swallow one teaspoon of applesauce
* Ask patient to chew one cracker

The following outcomes will be measured in both evaluations:

* Timing of swallow onset (timing of hyoid elevation)
* Duration of pharyngeal phase of swallow
* Timing of esophageal phase onset
* Duration of esophageal phase of swallow
* Coughing (Yes/No)
* Throat clearing (Yes/No)
* Pharyngeal pooling (Yes/No)
* Spontaneous multiple swallows (more than one) to clear bolus (Yes/No)

The investigator will compare the data obtained using videofluoroscopy swallowing study with the signals recorded with the electronic stethoscope to determine whether the patterns detected by electronic stethoscope concur with those obtained via the videofluoroscopy swallowing study. Additionally, the investigator will compare the results to similar tests performed by nurses and swallowing therapists.

Lastly, the investigators will compare the data obtained by the electronic stethoscope from the healthy controls in Phase I with the data obtained from the stroke patients in Phase II, and the investigators will try to determine whether the signals recorded can differentiate normal from abnormal swallowing patterns.

Patients will not be compensated for their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to CSMC for acute ischemic or hemorrhagic stroke, or TIA
2. No history of head and/or neck cancer
3. No tracheostomy or ventilator
4. Able to follow simple one step commands
5. 18 years of age or older

Exclusion Criteria:

1. Not admitted to CSMC for acute ischemic or hemorrhagic stroke or TIA
2. History of head and/or neck cancer
3. Tracheostomy or ventilator
4. Unable to follow simple one step commands
5. Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase 1: Normal Controls
  Phase 2: Patients with new onset Ischemic, hemorrhagic or transient ischemic attack
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Acoustic Signal of Normal Swallowing Pattern | 1 minute
  To establish the acoustic signals associated wtih a normal pattern of swallowing using an electronic stethoscope
Acoustic Signal of Swallowing in the Stroke Population | 1 minute
  To establish the acoustic signals associated with neurologic pattern of swallowing using an electronic stethoscope

IPD SHARING:
Plan to Share IPD: No
Data will only be shared in the aggregate

REFERENCES:
- [Background] Armstrong JR, Mosher BD. Aspiration pneumonia after stroke: intervention and prevention. Neurohospitalist. 2011 Apr;1(2):85-93. doi: 10.1177/1941875210395775. PMID 23983842
- [Background] Bhattacharyya N. The prevalence of dysphagia among adults in the United States. Otolaryngol Head Neck Surg. 2014 Nov;151(5):765-9. doi: 10.1177/0194599814549156. Epub 2014 Sep 5. PMID 25193514
- [Background] Brogan E, Langdon C, Brookes K, Budgeon C, Blacker D. Dysphagia and factors associated with respiratory infections in the first week post stroke. Neuroepidemiology. 2014;43(2):140-4. doi: 10.1159/000366423. Epub 2014 Nov 5. PMID 25402187
- [Background] Daniels SK, Brailey K, Priestly DH, Herrington LR, Weisberg LA, Foundas AL. Aspiration in patients with acute stroke. Arch Phys Med Rehabil. 1998 Jan;79(1):14-9. doi: 10.1016/s0003-9993(98)90200-3. PMID 9440410
- [Background] Edmiaston J, Connor LT, Steger-May K, Ford AL. A simple bedside stroke dysphagia screen, validated against videofluoroscopy, detects dysphagia and aspiration with high sensitivity. J Stroke Cerebrovasc Dis. 2014 Apr;23(4):712-6. doi: 10.1016/j.jstrokecerebrovasdis.2013.06.030. Epub 2013 Jul 30. PMID 23910514
- [Background] Kendall KA, McKenzie S, Leonard RJ, Goncalves MI, Walker A. Timing of events in normal swallowing: a videofluoroscopic study. Dysphagia. 2000 Spring;15(2):74-83. doi: 10.1007/s004550010004. PMID 10758189
- [Background] Leder SB, Bayar S, Sasaki CT, Salem RR. Fiberoptic endoscopic evaluation of swallowing in assessing aspiration after transhiatal esophagectomy. J Am Coll Surg. 2007 Oct;205(4):581-5. doi: 10.1016/j.jamcollsurg.2007.05.027. PMID 17903733
- [Background] Trapl M, Enderle P, Nowotny M, Teuschl Y, Matz K, Dachenhausen A, Brainin M. Dysphagia bedside screening for acute-stroke patients: the Gugging Swallowing Screen. Stroke. 2007 Nov;38(11):2948-52. doi: 10.1161/STROKEAHA.107.483933. Epub 2007 Sep 20. PMID 17885261